CLINICAL TRIAL: NCT03478176
Title: Intraabdominal Hypertension After Kidney Transplantation : Incidence and Associated Factors
Brief Title: Intraabdominal Hypertension After Kidney Transplantation
Acronym: KITIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PZ17048
Record Dates: First submitted 2018-02-01; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Intraabdominal Hypertension; Kidney Transplantation
Keywords: Intraabdominal hypertension; Kidney transplantation
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients

SUMMARY:
Intraabdominal hypertension (IAH) is a frequent and severe condition affecting intensive care patients. Gold standard for estimation of intraabdominal pressure is intravesical pressure (IVP) measurement. IVP measurement is recommended in patients presenting IAH risk factor(s). Acute kidney injury is the most frequent and described complication of IAH condition.

Patients undergoing kidney transplantation have several risk factors to develop IAH. Nevertheless, to our knowledge, IAH incidence, associated factors and impact on renal function recovery remains unknown.

We aim to study IAH incidence, associated factors and impact on renal function recovery in post kidney transplantation period.

DETAILED DESCRIPTION:
Intraabdominal hypertension (IAH) is a frequent and severe condition affecting 30 to 54% of intensive care patients. Gold standard for estimation of intraabdominal pressure is intravesical pressure (IVP) measurement. IAH is defined by IVP elevation above 12mmHg. IVP measurement is recommended in patients presenting IAH risk factor(s). Acute kidney injury (AKI)is the most frequent and described complication of IAH condition. IAH related AKI traduces renal hypoperfusion and its severity seems to correlate with IVP levels.

Patients undergoing kidney transplantation have several risk factors to develop IAH : abdominal wall surgery, acidosis and hypervolemic resuscitation. Nevertheless, to our knowledge, IAH incidence, associated factors and impact on renal function recovery remains unknown.

We aim to study IAH incidence in post kidney transplantation period. Thus, we want to identify associated factors with IAH development in this context. We also aim to correlate IVP early evolution with extra-cellular hydration status evolution. Finally, impact of IAH on renal function recovery will be investigated.

Presupposing that 50 kidney transplantations per year will take place in University Hospital of Reims (France), we attend to include about 100 patients in this study. With a prevalence of at least 30% of IAH prevalence (as reported in intensive care units cohorts), enrollment of 100 patients will permit to estimate IAH prevalence with a 9% precision (with a 95%IC).

ELIGIBILITY:
Inclusion Criteria:

* End stage chronic kidney disease ;
* Hospitalized in intensive care of nephrology unit in University Hospital of Reims (France) during study period ;
* Undergoing kidney transplantation ;
* Accepting to participate.

Exclusion Criteria:

* Minor ;
* Protected by the law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease undergoing kidney transplantation in University Hospital of Reims (France)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-05-08 (Estimated); Study Completion 2019-11-08 (Estimated)

PRIMARY OUTCOMES:
Intraabdominal hypertension Intraabdominal pressure | day 5
  Intraabdominal pressure equal or more than 12 mmHg for at least 2 measures spaced less than 24 hours. Intraabdominal pressure will be evaluated every 8 hours during the 5 days after transplantation, using UnometerTM AbdopressureTM system

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Derived] Dupont V, Debrumetz A, Leguillou A, Morland D, Wynckel A, Colosio C, Mokri L, Schvartz B, Vuiblet V, Larre S, Barbe C, Rieu P. Intra-abdominal hypertension in early post-kidney transplantation period is associated with impaired graft function. Nephrol Dial Transplant. 2020 Sep 1;35(9):1619-1628. doi: 10.1093/ndt/gfaa104. PMID 32678426